CLINICAL TRIAL: NCT01726478
Title: Uterotonic Efficacy of Oxytocin 2.5 Versus 10 Units During Caesarean Section at Mulago Hospital; Adouble Blinded Clinical Trial.
Brief Title: Uterotonic Efficacy of Oxytocin 2.5 Versus 10 Units During Caesarean Section at Mulago Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine (Other)
Responsible Party: Sponsor-Investigator, Faculty of Medicine, Dr Andrew Kintu, Makerere University
Organization: Makerere University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXY168
Record Dates: First submitted 2012-11-03; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Adverse Effect of Oxytocic Drugs; Uterine Hemorrhage; Inappropriate Dose of Drug Administered
Keywords: Oxytocin; Uterine tone; Mulago Hospital; Dose; Side effects
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2.5 units oxytocin (Active Comparator): Administration of 2.5 units of oxytocin intravenously after clamping of umbilical cord
  Interventions: Drug: 2.5 units Oxytocin
- 10 units oxytocin (Placebo Comparator): Administration of 10 units of oxytocin after clamping of umbilical cord
  Interventions: Drug: 10 units Oxytocin

INTERVENTIONS:
Drug: 2.5 units Oxytocin — Administration of 2.5 units of oxytocin after clamping of umbilical cord
  Other Names: pitocin
  Arms: 2.5 units oxytocin
Drug: 10 units Oxytocin — Administration of 10 units of oxytocin after clamping of umbilical cord
  Other Names: pitocin
  Arms: 10 units oxytocin

SUMMARY:
The purpose of the study was to determine whether 2.5 international units of oxytocin gives adequate uterine tone and is safe as compared to 10 international units of oxytocin following caesarean section delivery at Mulago hospital.

ELIGIBILITY:
Inclusion Criteria:

* ASA I (Healthy patient with no systemic disease) or II ( mild to moderate systemic disease)
* Age between 18 to 40 years
* Singleton pregnancies

Exclusion Criteria:

* • Allergy to oxytocin

  * Ruptured uterus
  * Significant obstetric disease (including Pregnancy induced Hypertension, Eclampsia,)
  * Known risk factors for postpartum haemorrhage or uterine atony
  * Inherited or acquired coagulation disorder
  * History of post partum haemorrhage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 386 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Uterine tone adequacy | 2 minutes
  The primary outcome was the assessment of either adequate or inadequate Uterine tone at various times after administration of initial oxytocin dose

SECONDARY OUTCOMES:
Intraoperative blood loss | 24 hours
  Blood loss was estimated by measuring the amount in the suction bottles and weighing of the mops. The patients were followed up for any occurrence of postpartum haemorrhage for the next 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kintu, MBChB, Principal Investigator — Makerere University College of Health Sciences Department of Anaesthesia
Locations (1):
- Mulago Hospital Labour Suite Operating Theatres, Kampala, East Africa, Uganda